CLINICAL TRIAL: NCT06171308
Title: Effect of Moxibustion Intervention on Insomnia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-YJ14
Record Dates: First submitted 2023-10-18; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-10

CONDITIONS: Insomnia; Moxibustion
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group(using the moxibustion) (Active Comparator): The study group was treated with traditional Chinese moxibustion and western medicine. The control group was treated with blank moxibustion and western medicine.
  1. The study group: Using the moxibustion, select specific 3 groups of acupoints. Select a group of acupuncture points every day, in the moxibustion treatment for 20 minutes, 4 weeks for a course of treatment.
  2. The control group: Using the moxibustion with blank patch, select specific 3 groups of acupoints. Select a group of acupuncture points every day, in the moxibustion treatment for 20 minutes, 4 weeks for a course of treatment.
  3. The treatment period is 4 weeks, which is a course of treatment, and the observation period is 8 weeks.
  Interventions: Device: Traditional Chinese moxibustion apparatus
- The control group(using the moxibustion with blank patch) (Placebo Comparator): The study group was treated with traditional Chinese moxibustion and western medicine. The control group was treated with blank moxibustion and western medicine.
  1. The study group: Using the moxibustion, select specific 3 groups of acupoints. Select a group of acupuncture points every day, in the moxibustion treatment for 20 minutes, 4 weeks for a course of treatment.
  2. The control group: Using the moxibustion with blank patch, select specific 3 groups of acupoints. Select a group of acupuncture points every day, in the moxibustion treatment for 20 minutes, 4 weeks for a course of treatment.
  3. The treatment period is 4 weeks, which is a course of treatment, and the observation period is 8 weeks.
  Interventions: Device: Traditional Chinese moxibustion apparatus

INTERVENTIONS:
Device: Traditional Chinese moxibustion apparatus — The study group was treated with traditional Chinese moxibustion and western medicine. The control group was treated with blank moxibustion and western medicine.
  1. The study group: Using the moxibustion, select specific 3 groups of acupoints. Select a group of acupuncture points every day, in the moxibustion treatment for 20 minutes, 4 weeks for a course of treatment.
  2. The control group: Using the moxibustion with blank patch, select specific 3 groups of acupoints. Select a group of acupuncture points every day, in the moxibustion treatment for 20 minutes, 4 weeks for a course of treatment.
  3. The treatment period is 4 weeks, which is a course of treatment, and the observation period is 8 weeks.

SUMMARY:
Type of study:clinical trial Purpose of research:To explore the efficacy and safety of moxibustion combined with Traditional Chinese and Western medicine in treating insomnia.

Describe participant population/health conditions:120 insomnia patients

DETAILED DESCRIPTION:
Type of study:clinical trial Purpose of research:To explore the efficacy and safety of moxibustion combined with Traditional Chinese and Western medicine in treating insomnia.

Describe participant population/health conditions:120 insomnia patients The participants were enrolled according to the principle of randomization and single blindness, and the analysis was adjusted every quarter according to the research schedule. The study group was treated with traditional Chinese moxibustion and western medicine. The control group was treated with only western medicine.

Clinical evaluation of the main efficacy indicators: The score of PSQI scale was assessed. The reduction rate of PSQI scale was ≥ 25% as effective, and the difference between the two groups was compared as the basis for evaluating the main efficacy indicators. The efficacy of insomnia symptoms was evaluated by the difference of PSQI score reduction rate between groups before and after intervention.

Secondary clinical outcome measures: Quality of Life Scale (SQLS), SF-36 scale, Clinical Gross Impression Scale (CGI), adverse reaction（TESS） .

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria of ICD-10 insomnia;
2. In line with the relevant diagnostic criteria of TCM syndrome differentiation of heart-spleen and deficiency type insomnia (TCM syndrome diagnosis criteria according to the 1993 Ministry of Health "Guidelines for Clinical Research on the treatment of Insomnia with new Chinese Medicine" standards: heart-spleen and deficiency: palpitation, amnesia, dizziness, poor and tired, pale face, easy to sweat, tongue, thin coat, thin pulse);
3. Pittsburgh Sleep Quality Index (PSQI) score > 7 at baseline;
4. The treatment plan used in this study is tolerable, cooperative and compliant;
5. Regardless of gender, age 18-65 years old;
6. Understand the procedure and content of the test, and voluntarily sign the informed consent;

Exclusion Criteria:

1. Participating in other clinical studies;
2. Exclude patients with serious physical diseases or diseases that may affect the evaluation of the test;
3. there is a clear risk of suicide or danger to oneself or others;
4. Exclude pregnant or lactating women, or those planning pregnancy;
5. Persons with alcohol and drug dependence within 1 year prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The score of PSQI | Baseline, week two, week four, week eight
  The reduction rate of PSQI scale ≥25% was regarded as effective, and the difference between the two groups was compared as the basis for evaluating the main therapeutic effect indicators. The efficacy of insomnia symptoms was evaluated by the difference in the reduction rate of PSQI scores between the two groups before and after the intervention.

SECONDARY OUTCOMES:
The score of Quality of Life Scale (SQLS) | Baseline, week two, week four, week eight
  The score reduction rate was taken as the therapeutic grade standard, and the score reduction rate =[(pre-treatment score - post-treatment score) ÷ pre-treatment score]×100%. The score reduction rate after treatment was ≥ 75% for clinical recovery, 50%-75% for obvious effect, 25%-50% for effective, and < 25% for ineffective. Total response rate = (effective + effective + cured)/total cases *100%.
The score of SF-36 scale | Baseline, week two, week four, week eight
  The score reduction rate was taken as the therapeutic grade standard, and the score reduction rate =[(pre-treatment score - post-treatment score) ÷ pre-treatment score]×100%. The score reduction rate after treatment was ≥ 75% for clinical recovery, 50%-75% for obvious effect, 25%-50% for effective, and < 25% for ineffective. Total response rate = (effective + effective + cured)/total cases *100%.
The score of Clinical Gross Impression Scale (CGI) | Baseline, week two, week four, week eight
  The score reduction rate was taken as the therapeutic grade standard, and the score reduction rate =[(pre-treatment score - post-treatment score) ÷ pre-treatment score]×100%. The score reduction rate after treatment was ≥ 75% for clinical recovery, 50%-75% for obvious effect, 25%-50% for effective, and < 25% for ineffective. Total response rate = (effective + effective + cured)/total cases *100%.
adverse reaction（TESS）evaluation | Baseline, week two, week four, week eight
  The score reduction rate was taken as the therapeutic grade standard, and the score reduction rate =[(pre-treatment score - post-treatment score) ÷ pre-treatment score]×100%. The score reduction rate after treatment was ≥ 75% for clinical recovery, 50%-75% for obvious effect, 25%-50% for effective, and < 25% for ineffective. Total response rate = (effective + effective + cured)/total cases *100%.

CONTACTS AND LOCATIONS:
Locations (1):
- moxibustion equipment（Zhongshan Jiaxun medical equipment Co., LTD）, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No